CLINICAL TRIAL: NCT00386542
Title: Clinical Trial of Safety (Reactogenicity) and Immunogenicity of Needle-free Jet Injection of Reduced-dose, Intradermal Influenza Vaccine (INF) Administered to >= 6 to < 24 Month-old Infants and Toddlers in the Dominican Republic
Brief Title: Needle-free Jet Injection of Reduced-dose, Intradermal, Influenza Vaccine in >= 6 to < 24-month-old Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pedro Moro (U.S. Federal Agency)
Collaborators: Fundación Dominicana de Infectología, Santo Domingo, Dominican Republic (Unknown); Hospital Infantil Dr. Robert Reid Cabral (Other); World Health Organization (Other); Pan American Health Organization (Other); PATH (Other); Bioject Medical Technologies, Inc. (Industry); MCM Vaccines B.V. (Industry)
Responsible Party: Sponsor-Investigator, Pedro Moro, epidemiologist, Centers for Disease Control and Prevention
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDC-ISO-4785
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Influenza
Keywords: vaccination; influenza vaccine; jet injection; intradermal injection; infancy; children; dose-sparing; cutaneous vaccination; Dominican Republic; pandemic preparedness; jet injector; reduced dosage; immunogenicity; reactogenicity; safety; needle-free; immune response; hemagglutination inhibition; Infant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ID-JI-0.1 (Experimental): Group "ID-JI-0.1" (n = 16) - reduced 0.1 mL INF doses administered intradermally (ID) by needle-free jet injector (JI) (Biojector® 2000 subcutaneous syringe no. 2 [green color code], with 2 cm investigational spacer, Bioject Medical Technologies, Inc., Portland, OR, USA)
  Interventions: Biological: Vaxigrip® trivalent inactivated influenza vaccine; Device: Intradermal spacer on Biojector® 2000 jet injector
- IM-NS-0.1 (Active Comparator): Group "IM-NS-0.1" (n = 16) - reduced 0.1 mL INF doses administered intramuscularly (IM) needle-syringe (NS) (via 22-25 gauge needle, minimum 25 mm/1-inch length)
  Interventions: Biological: Vaxigrip® trivalent inactivated influenza vaccine
- IM-NS-0.25 control (Active Comparator): Group "IM-NS-0.25" (controls) (n = 16) - full 0.25 mL INF doses administered intramuscularly (IM) by needle-syringe (NS) (22-25 gauge needle, minimum 25 mm/1-inch length)
  Interventions: Biological: Vaxigrip® trivalent inactivated influenza vaccine

INTERVENTIONS:
Biological: Vaxigrip® trivalent inactivated influenza vaccine — See full description elsewhere in this record.
Device: Intradermal spacer on Biojector® 2000 jet injector — See elsewhere in this record for full description.
  Arms: ID-JI-0.1

SUMMARY:
This is a sequential phase I and II, controlled, double-blinded study to determine whether immune responses suggesting protection against influenza can safely be induced in young children by two reduced doses one month apart of 0.1 mL of a trivalent inactivated influenza vaccine (INF) administered by the intradermal (ID) route with an investigational ID spacer on a United States (U.S.)-licensed needle-free jet injector (JI), compared to two standard intramuscular (IM) 0.25 mL doses by needle-syringe (N-S) in this age group. The locale is a developing country where financial restraints for the use of full-dose influenza vaccine would limit protection from an influenza pandemic threat, where N-Ss pose dangers and drawbacks in clinical use, and where Mantoux-type N-S ID injections are difficult to administer during mass campaigns.

DETAILED DESCRIPTION:
Randomized, observer-blinded, clinical pilot (phase I) trial of safety, followed by a clinical (phase II) trial of safety and non-inferiority of immune response to the standard route and dose for the merged subjects from both phases.

Phase I - Influenza-vaccine naïve children (n = 48) aged >= 6 to < 24 months will be randomized in a 1:1:1 ratio to the following three study arms, each to receive two doses on days 0 and 28 of trivalent inactivated influenza (INF) vaccine (Vaxigrip®, Sanofi Pasteur, Lyon, France) into the left thigh (< 12 months) or left deltoid (≥ 12 months):

* Group "ID-JI-0.1" (n = 16) - reduced 0.1 mL INF doses administered intradermally (ID) by needle-free jet injector (JI) (Biojector® 2000 subcutaneous syringe no. 2 [green color code], with 2 cm investigational spacer, Bioject Medical Technologies, Inc., Portland, OR, USA)
* Group "IM-NS-0.1" (n = 16) - reduced 0.1 mL INF doses administered intramuscularly (IM) needle-syringe (NS) (via 22-25 gauge needle, minimum 25 mm/1-inch length)
* Group "IM-NS-0.25" (controls) (n = 16) - full 0.25 mL INF doses administered intramuscularly (IM) by needle-syringe (NS) (22-25 gauge needle, minimum 25 mm/1-inch length)

Phase II - Upon assessment of the safety profile from phase I by the unblinded Data Safety Monitoring Board (DSMB), with its approval an additional 402 children will be recruited and randomized (134 per group) as in phase I above. Total subjects in phase I and II = 450 (150 in each of three study arms).

Adverse Event Diaries: Parents will be trained to complete a diary form to observe, measure, and record solicited local reactions for the injection site and systemic signs and symptoms for the child for days 0 through 7 after vaccination, plus unsolicited symptoms, illness, and medications for days 0 through 28.

Followup: Return clinic visits will be scheduled on days 2, 7, and 28 after INF dose 1, at which times the diary card data will be recorded by staff and the card collected on day 28. Upon receiving dose 2 of vaccine, patients will be scheduled again to return to the study center 2, 7, and 28 days afterwards. The same procedures as for dose 1 regarding diary cards, telephone followup, and home visits will apply after dose 2.

Upon returning to clinic on day 28 after dose 2 (day 56 after dose 1), the child will receive an unblinded, "insurance", full-volume, 0.25 mL dose (#3) of influenza vaccine by NS IM, unless he or she is in the full-dose IM control group IM-NS-0.25, in which case a mock injection will be administered instead of a 3rd full dose beyond the usual 2-dose series. All participants will return 6 months after this third injection for a fourth "bonus" dose of influenza vaccine to ensure protection for the following season.

Serum Collection: Blood specimens to measure serologic responses will be collected three times, just prior to vaccination on day 0 (INF dose 1), on day 28 (INF dose 2), and on day 56 (INF "insurance" dose 3).

Ethical oversight additional to CDC IRB G by (1) World Health Organization Research Ethics Review Committee, (2) Consejo Nacional de Bioética en Salud, and (3) Fundación Dominicana de Infectología Comité de Etica/Investigaciones.

ELIGIBILITY:
Inclusion Criteria:

* Age from > = 6 to < 24 months (not having reached 2nd birthday).
* Born after a full-term (≥ 37 weeks), and birth weight of >= 2.5 kg (>= 5 pounds, 8 ounces)
* History of prior or first attendance as a patient, or as a sibling of a patient, seeking routine immunization or other clinical care at the Hospital Infantíl Robert Reid Cabral (HIRRC)
* The parent(s) or legal guardian(s) provide(s) written informed consent and agree(s) to bring the infant back to the clinic for all visits scheduled in the study
* Up-to-date for routine doses of vaccines officially recommended for the patient's age in the Dominican Republic to prevent tuberculosis, polio, diphtheria, tetanus, pertussis, hepatitis B, and Haemophilus influenzae B
* In good health, as determined by medical history and physical examination collected in accordance with the Case Report Form (CRF), and by the clinical judgment of the investigators.

Exclusion Criteria:

Infants WHOSE PARENT(S)/LEGAL GUARDIAN(S):

* Are unable or unwilling to give written informed consent for their infant to participate in the study
* Cannot be contacted by telephone (family's own or a neighbor's) if necessary for adverse events if scheduled followup return appointments are missed
* Are unable to complete the diary for adverse events; are unable to measure and record temperatures or maximal diameter of local reactions or limb circumference; or have difficulty understanding written instructions; or other factors which indicate exclusion in the judgement of the study staff.

INFANTS who:

* Have fever (by parental report or by rectal temperature ≥ 38.5° C or axillary ≥ 38.0° C) currently or within the past 3 days, or who are currently suffering from an acute or chronic infectious disease (including known HIV)
* Have had an acute or chronic infection requiring systemic antimicrobial therapy (antibiotic or antiviral) or other prescribed treatment within the past 21 days. This includes any underlying illness that may limit their response to vaccination, such as those receiving intravenous immunoglobulin for agammaglobulinemia, or systemic steroid therapy.
* Are malnourished, defined by weight less than two standard deviations below the median weight for their age
* Are allergic to eggs, or have a history of any anaphylactic shock, asthma, urticaria, or other allergic reaction after previous vaccinations, or have allergy or hypersensitivity to any component of the study vaccine
* Have ever previously received any influenza vaccine
* Have received within the prior 28 days, or for whom there is the indication to receive in the next 56 days, any non-study vaccination or investigational agent outside of the study
* Have a known bleeding diathesis, or any condition with a prolonged bleeding time
* Currently have any serious confirmed or suspected disease, such as metabolic, cardiac, or autoimmune disease, or diabetes
* Have a history of epilepsy or a seizure disorder, or neurodevelopmental disorders such as autism
* Have a genetic anomaly or known cytogenic disorder (e.g., Down's syndrome)
* Have leukemia, lymphoma, or any other cancer/neoplasm
* Have known or suspected immune dysfunction, including HIV infection, or receives(ed) immunosuppressive therapy, including systemic corticosteroids
* Have ever received blood, blood products, or parenteral preparations of immunoglobulin
* Have any other serious disease (e.g., with signs of cardiac or renal failure), including progressive neurologic disease
* Have any condition which, in the opinion of the investigator, may interfere in the evaluation of the objectives of the study

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2006-10; Primary Completion 2009-11 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Rates of seroconversion (SC) on HI assay 1 month after dose 2. SC defined as titer >= 40 among initial-seronegatives (titer < 8 on day 0); OR, a followup titer which rises >= 4-fold. | One month after each of doses 1 and 2.
  seroconversion and safety assessed through occurrence of local and systemic reactions

SECONDARY OUTCOMES:
Rates of local and systemic reactions | Up to 42 days for prompted symptoms after investigational doses 1 and 2. Up to 6 months for unsolicited ones.
  assessment of these reactions by study investigators
Seroprotection (SP) on HI assay, defined as >= 40 regardless of baseline | One month after each of doses 1 and 2.
  assays were performed at CDC
Geometric mean titers (GMT) on HI | One month after each of doses 1 and 2.
  assays were performed at CDC
Geometric mean increase (GMI) on HI | One month after each of doses 1 and 2.
  assays were performed at CDC

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G Weniger, MD, MPH, Principal Investigator — CDC (bgweniger@siamlotus.com) (bgw2@cdc.gov obsolete by 2021).com); Virgen Gómez, MD, Study Director — Hospital Infantíl Dr. Robert Reid Cabral; Jesús M Feris Iglesias, MD, Study Director — Hospital Infantíl Dr. Robert Reid Cabral; Josefina Fernández, MD, Study Director — Hospital Infantíl Dr. Robert Reid Cabral; Pedro Moro, MD, MPH, Study Director — Immunization Safety Office, Centers for Disease Control and Prevention; Martin Friede, PhD, Study Chair — Initiative for Vaccine Research, World Health Organization
Locations (1):
- Hospital Infantíl Dr. Robert Reid Cabral, Santo Domingo, Nacional, Dominican Republic

REFERENCES:
- [Result] Palomeque FS, Weniger BG, Jet-Injected Cutaneous Influenza Vaccination Study Group. History and Technologies for Cutaneous Influenza Vaccination; and Preliminary Results from a CDC Trial of Jet-Injected, Needle-free Influenza Vaccine in ≥6 to <24-month-old Children in the Dominican Republic. CDC Vaccine Technology Seminar Series & CDC Influenza Division Seminar Series (Centers for Disease Control and Prevention), Atlanta, GA, 24 September 2013
- See also: Palomeque FS, Weniger BG, Jet-Injected Cutaneous Influenza Vacc. Study Group. Hist. & Technol. Cutaneous Influenza Vaccin.; & Prelim. Results CDC Trial Jet-Injected, Needle-free Infl. Vacc. ≥6-<24-mos-olds in Dom. Rep. (CDC Presentation) — https://bit.ly/Cutaneous-influenza-vacc-trial
- Available data/document: Interim results presentation — https://web.archive.org/web/20210528232541/https://siamlotus.com/ppt-2013-meetingpresentations/Palomeque&Weniger_History-Cutaneous-Influenza+Trial-Results_CDC-Atlanta_2013-09-24_Color-handouts.pdf — Palomeque FS, Weniger BG, Jet-Injected Cutaneous Influenza Vaccination Study Group. History and Technologies for Cutaneous Influenza Vaccination; and Preliminary Results from a CDC Trial of Jet-Injected, Needle-free Influenza Vaccine in ≥6 to <24-month-old Children in the Dominican Republic. CDC Vaccine Technology Seminar Series & CDC Influenza Division Seminar Series (Centers for Disease Control and Prevention), Atlanta, GA, 24 September 2013

DOCUMENTS (2):
  • Study Protocol (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT00386542/Prot_000.pdf
  • Informed Consent Form (2007-03-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT00386542/ICF_001.pdf